CLINICAL TRIAL: NCT01058538
Title: A Dose Finding Pharmacokinetic Study of the Tumour-targeting Human L19IL2 Monoclonal Antibody-Cytokine Fusion Protein in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2-01/05; 2005-002716-16 (EudraCT Number)
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Solid Tumours
Keywords: Interleukin, IL2, monoclonal, antibody, cytokine, tumour targeting, solid tumours, dose finding, renal cell carcinoma, fusion protein, RCC,; L19
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L19IL2 (Experimental)
  Interventions: Drug: L19IL2

INTERVENTIONS:
Drug: L19IL2 — Route: i.v. infusion (60 min) Patients will receive a minimum of 2 cycles of treatment. Each cycle is comprised of treatment on Days 1, 3 and 5 followed by a 16 days rest (1 cycle= 21 days). Patients may receive up to 4 further cycles of treatment (max. of 6 cycles in total). Patients will be initially recruited into the study in cohorts of 3 and the starting dose of L19IL2 will be 5 Mio IU IL2 equivalent. Five steps of dose escalation are planned: 5, 10, 20, 30 and 40 Mio IU IL2 equivalent). After the MTD has been established, the RD will be determined. A further 12 patients (with RCC) will receive the RD dose for a minimum of 2 cycles. For patients in the RD part of the study, patients can switch to maintenance therapy. Maintenance therapy consists of 15 Mio IU IL2 every 2 weeks. The maximum duration of the study for a patient is 12 months.

SUMMARY:
This is a Phase I/II study for patients with solid tumors and renal cell carcinoma (RCC; for the Phase II part). L19-IL2 is a tumor targeted immunocytokine constituted of a single chain Fragment variable (scFv) format directed against the ED-B domain of fibronectin, one of the most important markers for neoangiogenesis, and the human cytokine interleukin-2 (IL2).

DETAILED DESCRIPTION:
This is an open-label, non-randomised, multicentre, Phase I/II study to assess safety, pharmacokinetics (PK), and early signs of activity of L19-IL2 monotherapy.

In the first part of the study, there will be 5 dose escalation steps in sequential cohorts of patients with advanced solid tumours. In the second part of the study, patients with advanced RCC will be given a fixed dose of L19IL2 at the RD.

ELIGIBILITY:
Inclusion Criteria:

* For the first part of the study: histologically or cytologically confirmed solid cancer with evidence of advanced disease for which no other standard treatment is available or appropriate. For the second part of the study: Histologically or cytologically confirmed advanced RCC.
* Patients must have at least one measurable lesion as detected by computed tomography (CT).
* All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v3.0) Grade </=1.
* Patients who have received autologous marrow/stem cell infusion using monoclonal antibody-purged specimens are eligible.
* Adult patients of both sexes aged 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status </=2.
* Sufficient haematological, liver and renal function:
* Absolute neutrophil count (ANC) >/=1.5 x 109/L, platelets >/=100 x 109/L, haemoglobin (Hb) >/=9.0 g/dL,
* Alkaline phosphatase (AP) </=3 x upper limit of the reference range (ULN) and alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) </=3 x ULN, and bilirubin <1.5 x ULN; however, in the presence of liver metastases, AP </=5 x ULN and ALT and/or AST </=5 x ULN, and bilirubin <1.5 x ULN,
* Creatinine </=ULN, or 24 h creatinine clearance >/=50 mL/min.
* Pulse oximetry >94% on room air.
* Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment.
* Life expectancy of at least 3 months.
* Evidence of a personally signed and dated informed consent indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.
* Negative human immunodeficiency virus (HIV) test 2 to 3 weeks before administration of study treatment (with informed consent for test taken).

Exclusion Criteria:

* Presence of active infections (eg requiring antibiotic therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* Presence of known brain metastases.
* Chronic aggressive hepatitis or active autoimmune diseases.
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
* Heart insufficiency (>Grade II New York Heart Association [NYHA] criteria).
* Irreversible cardiac arrhythmias requiring permanent medication.
* Uncontrolled hypertension.
* Ischaemic peripheral vascular disease (Grade IIb-IV).
* Severe rheumatoid arthritis.
* Severe diabetic retinopathy.
* Recovery from major trauma including surgery within 4 weeks of administration of study treatment.
* Known history of allergy to intravenously administered proteins/peptides/antibodies.
* Pregnancy or breast feeding. Female patients must agree to use effective contraception, or be surgically sterile or postmenopausal. The definition of effective contraception will be based on the judgement of the principal investigator or a designated associate.
* Chemotherapy (standard or experimental) within 4 weeks of the administration of study treatment, or 6 weeks for nitrous ureas, l-phenylalanine mustard (LPAM) or temozolamide.
* Radiation therapy within 4 weeks of the administration of study treatment.
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment.
* Growth factors or immunomodulatory agents within 7 days of the administration of study treatment.
* Prior allografts (including bone marrow or stem cells).
* Patient requires or is taking corticosteroids or other immunosuppressant drugs on a long term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
* Investigational study drug taken within 4 weeks of the administration of study treatment or concurrent treatment with other anti-cancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and recommended dose (RD) of the human L19IL2 fusion-cytokine. | 21 days

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile. | 5 days
To determine the qualitative and quantitative toxicity profile. | 21 days
To assess the presence of anti-fusion protein antibodies in treated patients. | 18 weeks
To evaluate the safety profile of repeated administrations of L19IL2 in patients treated at the RD. | 1 year
To identify early signs of antitumour activity. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Filippo De Braud, Dr, Principal Investigator — European Institute of Oncology Milan (Italy); Manfred Johannsen, Dr, Principal Investigator — Champus Charitè Mitte Berlin (Germany)
Locations (2):
- Campus Charité Mitte, Berlin, Germany
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Johannsen M, Spitaleri G, Curigliano G, Roigas J, Weikert S, Kempkensteffen C, Roemer A, Kloeters C, Rogalla P, Pecher G, Miller K, Berndt A, Kosmehl H, Trachsel E, Kaspar M, Lovato V, Gonzalez-Iglesias R, Giovannoni L, Menssen HD, Neri D, de Braud F. The tumour-targeting human L19-IL2 immunocytokine: preclinical safety studies, phase I clinical trial in patients with solid tumours and expansion into patients with advanced renal cell carcinoma. Eur J Cancer. 2010 Nov;46(16):2926-35. doi: 10.1016/j.ejca.2010.07.033. Epub 2010 Aug 24. PMID 20797845